CLINICAL TRIAL: NCT05930769
Title: Retrospective Study on the Evaluation of the Impact of Augmented Reality Usage in Gynecological Laparoscopy on Patients Operated Between 2017 and 2021
Brief Title: Retrospective Study on the Evaluation of the Impact of Augmented Reality Usage in Gynecological Laparoscopy on Patients Operated Between 2017 and 2021 (ImpactRA)
Acronym: ImpactRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-CF016.
Record Dates: First submitted 2023-05-31; First posted 2023-07-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Myoma;Uterus; Adenomyoma of Uterus
Keywords: Augmented Reality; Uterine myomectomy; Uterine adenomyomectomy; Laparoscopic surgery; Minimally invasive surgery
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Patients that have undergone laparoscopy, with surgical indication of myomectomy or adenomyomectomy, with augmented reality (AR).
  Interventions: Procedure: Gynecological laparoscopic surgery with augmented reality
- Control group: Patients that have undergone laparoscopy, with surgical indication of myomectomy or adenomyomectomy, without augmented reality (AR).
  Interventions: Procedure: Gynecological laparoscopic surgery without augmented reality

INTERVENTIONS:
Procedure: Gynecological laparoscopic surgery without augmented reality — Minimally invasive gynecological surgery assisted by laparoscope.
  Groups: Control group
Procedure: Gynecological laparoscopic surgery with augmented reality — Minimally invasive gynecological surgery assisted by laparoscope with the display of additional information through augmented reality.
  Groups: Case group

SUMMARY:
ImpactRA is an observational retrospective study. The management of the patient is not modified by this study. This study will be carried out based on the already existing data of the gynecological ward of CHU Clermont-Ferrand between 2016 and 2021. During this period of time, 17 patients have undergone laparoscopy, with surgical indication of myomectomy or adenomyomectomy, aided by augmented reality (AR). The investigators compared these 17 patients that underwent surgery with AR with 17 control patients that underwent the same surgery with the same indication but without AR.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 (included) and 84 (Included),
* Patient operated between 2017* et 2021,
* Patient with one or more intrauterine myomas, with surgical treatment by laparoscopic myomectomy with or without AR,
* Patient with one or more intrauterine adenomyomas, with surgical treatment by laparoscopic adenomyomectomy with or without AR,
* Patient informed about the use of her data for research.

Exclusion Criteria:

* Patient who refused the use of medical data for research purposes,
* Patient operated prior to 2017* and after 2021,
* Patient whose medical follow-up did not allow collection of the data required for the study.

(*) An amendment validated by the ethics committee allows inclusion of patients operated during 2016

Ages: 18 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged between 18-84 years old that were indicated for an laparoscopic myomectomy or laparoscopic adenomyomectomy.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Operation duration (in minute) | In the intra-operative phase of the study
  Assessment of the use of augmented reality during gynecologic laparoscopy defined by the non-increase of the operation time.

SECONDARY OUTCOMES:
Amount of bleeding (in mL) | In the intra-operative phase of the study
  Estimating the impact of AR on the amount of bleeding
Post-operative pain measured with the visual analogue scale (VAS) score (measure every day after the operation as well as at the end of hospitalization). | In the post-operative phase of the study
  Estimating the impact of AR on the pain measured with the post-operative visual analogue scale (VAS) score. The score on this scale ranges from 0 to 10. The higher the score, the more pain the patient experienced at the time of filling in the scale.
Intra-operative complication number and details (wounds of adjacent structures and organs, vascular wounds, opening of the uterine cavity, difficulties in locating the tumor) based on the comments of the surgical report | In the intra-operative phase of the study
  Estimating the impact of AR on the intra-operative complication rate
Conversion from laparoscopy to laparotomy | In the intra-operative phase of the study
  Estimating the impact of AR on the conversion rate (laparoscopy to laparotomy)
Comments related to the set up of AR (according to the surgical report) | In the intra-operative phase of the study
  Estimating the impact of AR in the operating room represented by its installation and use during the course of the surgical procedure and estimating the impact of AR on the complexity/difficulty of the procedure recorded in the surgical report
Total time of hospitalization (in day) | From the date of hospital admission to the date of hospital discharge assessed up to 1 week
  Estimating the impact of AR on hospitalization duration
Time between discharge from hospital and the last post-operative visit (in months) | From the date of hospital discharge to the date of the latest post-operative visit, assessed up to the last available information for each specific patient (6 years)
  Estimating the impact of AR on the time between discharge from hospital and the last post-operative visit (in months)
Pregnancy obtention follow-up | From the date of surgery to the date of the latest post-operative visit, assessed up to the last available information for each specific patient (6 years)
  Estimating the impact of AR on the frequency of post-operative pregnancy
Adenomyosis / myoma(s) recurrence from 6 months after the operation ; | From the date of the surgery to the date of the latest post-operative visit, assessed up to the last available information for each specific patient (6 years)
  Estimating the impact of AR on the frequency of recurrence greater than 6 months
Post-operative complications numbers and details (wounds of adjacent structures and organs, bleeding complications, reoperations, complications based on the Clavien-Dindo classification) based on the comments of the post-operative consultation | From the date of the surgery to the date of the latest post-operative visit, assessed up to the last available information for each specific patient (6 years)
  Estimating the impact of AR on the post-operative complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Pauline CHAUVET, Principal Investigator — pchauvet@chu-clermontferrand.fr
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France